CLINICAL TRIAL: NCT06323252
Title: A Study on the Effects of Mastiha Oil in Adults With Hypertriglyceridemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Responsible Party: Principal Investigator, Andriana C Kaliora, Associate Professor in Foods and Human Nutrition, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MastihaOil-HT
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Participants with hypetriglyceridemia will be subjected to nutritional counsel and the intake of 1 soft gel capsule daily for a total of 3 months.
  Interventions: Dietary Supplement: MastihaOil
- Control group (Active Comparator): Participants with hypetriglyceridemia will be subjected to nutritional counsel for a total of 3 months.
  Interventions: Behavioral: nutritional counsel

INTERVENTIONS:
Dietary Supplement: MastihaOil — 1 soft gel capsule of Mastiha oil every day for 3 months
  Arms: Intervention group
Behavioral: nutritional counsel — nutritional counsel
  Arms: Control group

SUMMARY:
Mastiha Oil is a 100% natural product of the Mediterranean, extracted from the resin of Mastiha. Its composition is high in bioactive ingredients (such as terpenic acids and polyphenols) which have proven anti-inflammatory, antioxidant, cardioprotective, chemoprotective and antimicrobial properties. The aim of this study is to determine the effect of Mastiha oil in adults with Hypetriglyceridemia. 100 participants will be allocated to two groups, (50 in intervention group and 50 in control group). Mastiha oil will be provided in the form of soft gel capsules to the intervention group, whereas the control group will not consume the capsules. Both groups will receive standard nutritional counselling. The intervention will last 3 months.

The effects of the intervention will be evaluated via clinical and laboratory markers.

ELIGIBILITY:
Inclusion Criteria:

* 30 years < Age < 75 years Hypetriglyceridemia A stable weight for ≥ 3 months pre-intervention An unchanged treatment regimen for ≥ 6 months pre-intervention

Exclusion Criteria:

Hepatotoxic Medication Untreated Diabetes Mellitus Dysthyroidism, hypopituitarism, Cushing syndrome / disease Pregnancy, lactation Psychiatric or mental disorder Any use of antioxidant-phytochemical rich supplement, vitamin D supplement, anti-, pre- or pro-biotics within 3 months pre-intervention

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in blood triglycerides | 3 months
  Levels will be evaluated pre and prost intervention in both control and intervention groups

IPD SHARING:
Plan to Share IPD: Undecided